CLINICAL TRIAL: NCT05617365
Title: Treating Chronic Cervicogenic Head and Neck Pain With Osteopathic Manipulation and Exercise Therapy
Brief Title: Treating Chronic Cervicogenic Head and Neck Pain
Acronym: CGH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Richard Hallgren, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 016507-00001
Record Dates: First submitted 2022-11-05; First posted 2022-11-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cervicogenic Headache; Neck Pain, Posterior
MeSH Terms: conditions — Post-Traumatic Headache; Neck Pain | interventions — Manipulation, Osteopathic; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: The primary aim of our study is to test the combined effectiveness of osteopathic manipulative treatment (OMT) and targeted head exercise (THE) to achieve a significant decrease in headache measures of frequency, intensity, and duration in a Treatment group when compared to a Control group whose members receive only standard medical care.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): All subjects in the Treatment group will receive OMT a minimum 4 times and a maximum of 8 times at the physician's (JJR) discretion (Jull et al., 2002). All subjects in the Treatment group will be taught the THE. This voluntary head retraction/protrusion exercise protocol engages the RCPm muscles in eccentric and isometric contractions that should strengthen the muscles and thereby increase CSA.
  Interventions: Combination Product: Osteopathic Manipulative Therapy and Exercise Therapy
- Control (No Intervention): All subjects assigned to the Control group will be allowed to continue to receive conservative care. It is understood that any care that they receive will be prescribed on an individual basis. A participant could therefore receive any combination of medical, physio therapeutic and psychological care. It would also be expected that some form of pain management will be a priority for participants with moderate to severe symptoms. Subjects assigned to the Control group will not receive OMT and will not be taught the THE protocol.

INTERVENTIONS:
Combination Product: Osteopathic Manipulative Therapy and Exercise Therapy — At the physician's discretion, each subject will receive a minimum of 4 treatments up to a maximum of 8 treatments over the 12-week duration of the study (Haas et. al., 2018). The patients may be treated in the seated, prone and/or supine positions. Duration of treatment will depend on the degree of documented dysfunction but will be limited to one half hour. The techniques utilized by the physician may vary for many reasons including the degree of restriction, acuity, or patient cooperation.
  The THE protocol will involve subjects performing cyclic voluntary retraction and protrusion of their head.
  Arms: Treatment

SUMMARY:
The primary aim is to test the combined effectiveness of OMT and targeted head exercise (THE) to achieve a significant decrease in headache measures of frequency, intensity, and duration in a Treatment group when compared to a Control group whose members receive only standard medical care. A parallel, 2-arm, longitudinal, randomized controlled trial (RCT) will focus upon female patients (18 to 75 years of age) who have been diagnosed with chronic cervicogenic headache (CeH) based upon a differential diagnosis that includes classification according to the International Headache Society Classification IHSD 3rd Edition, reproduction of referred headache resulting from manual pressure over the upper cervical regions, and objective MRI findings. It is estimated that a sample size of 30 will provide sufficient statistical power (79%) to detect an intervention effect that corresponds to a clinically meaningful recovery (60%).

CeH is classified as a secondary headache disorder because the headache pain is a consequence of injury to, or disease of, the bony and/or soft tissues of the upper cervical spine. It has been reported that some patients diagnosed with CeH demonstrate atrophy and/or fatty infiltration (FI) of the RCPm muscles on MRI. FI and/or a reduction in the cross-sectional area (CSA) of active muscle would not be expected to be the direct cause of chronic headache, but either or both could prevent muscles from generating normal physiologic levels of force. It has been shown that there is a functional connection between the pain sensitive dura mater and RCPm muscles and it is known that mechanical stretching of the dura mater results in referred headache.

While FI and/or a reduction in the CSA of active muscle would not be expected to be the direct cause of chronic headache, it is known that muscle pathology will result in functional deficits. It is proposed that pathology in RCPm muscles will compromise the normal functional relationship between the RCPm and the dura mater and result in referred head and neck pain. It is predicted that at the end of the study, the Treatment group will show a significant decrease in headache measures that will be accompanied by a significant increase in CSA and a significant decrease in FI on MRI, and restoration of a normal head posture that will not be seen in the Control group.

The proposed study is unique in that we are proposing both a mechanism and a source for some instances of CeH. By testing the effectiveness of specific interventions to address a specific pathology within a specific headache population, and by restricting the study cohort to female subjects presenting with CeH, this study will increase the ability to detect a significant change in the outcomes by increasing the power of the statistical analysis.

DETAILED DESCRIPTION:
CeH preferentially effects female headache patients (Racicki et al., 2013). CeH is classified as a secondary headache disorder because the source of the pain is thought to be a consequence of injury to, or disease of, the bony and/or soft tissues of the upper cervical spine (Kristoffersen et al., 2017). Clinical management of CeH is challenging for the physician because a pathology that would account for the pain is usually unknown.

The primary diagnostic criteria that physicians use to diagnose CeH is based upon classification according to the International Headache Society Classification IHSD 3rd Edition (HIS, 2013). CeH is characterized by unilateral head or face pain without side shift that is of moderate to severe intensity of varying duration (Antonaci et al., 2001). CeH may occasionally be bilateral, throbbing, and accompanied by nausea, vomiting, phonophobia, photophobia, and dizziness when chronic tension-type headache and chronic migraine attacks are superimposed (Biondi, 2005). If the source of CeH originates in the upper cervical spine, osteopathic physicians can use head and neck movements and pressure applied to the suboccipital and lower cervical regions (Anarte-Lazo et al., 2021) to provoke referred headache. These diagnostic techniques, along with restricted active and passive range of motion (ROM) of the head and neck (Ogince et al., 2007), provide additional credibility that the diagnosis of CeH is valid (Avijgan et al., 2020) and helps ensure that the efficacy of our treatment protocol is not weakened by applying it to subjects with a different type of headache, such as migraine, that would not be expected to respond to a treatment protocol designed for CeH patients (Bogduk N, 2014).

The largest study of conservative therapy for cervicogenic headache (Jull et al., 2002) reported that manual therapy alone was not more effective than exercises alone. The study reported that headache frequency was reduced by 50% at a 7-week follow up, but figures for reduction in pain intensity were not reported. They reported that combining manipulation and exercise was not significantly superior to either therapy alone. Hidalgo et al., (2017) have reported that combining the 2 therapies is better than either manipulation or exercise alone. The weakness of Jull et al's. (2002) study was that their treatment protocol was applied to subjects who would not have had a common etiology for their headache pain. CeH is defined by injury to, or disease of, the bony and/or soft tissues of the upper cervical spine (Bogduk N, 2014). MRI is the gold standard for diagnostic assessment of structures of the upper cervical spine (Sun et al., 2020), but Jull et, al.'s (2002) study did not include an MRI assessment of the upper cervical spine in their inclusion/exclusion criteria. The outcome of their study reported that their treatment protocol showed a positive effect, but not one that rose to a significant level. I suggest this was due to mixing headache types (CM and CeH) that have different etiologies and expecting a single treatment protocol to address both pathologies.

Since CeH results from injury to, or disease of, the bony and/or soft tissues of the upper cervical spine, it is only reasonable to exclude those patients who do not present with pathology on MRI in the upper cervical spine (Sun et al.,2020). Our study is unique in that we will test the effectiveness of specific interventions that address a specific pathology within a specific headache population. By actively restricting the study cohort to a specific headache population, we will increase our ability to detect a significant change in the outcomes of treatment by increasing the power of the statistical analysis.

This study is unique in that it proposes to investigate a mechanism responsible for referred pain in some instances of chronic CeH. The effectiveness of specific interventions to address a specific pathology within a specific headache population will be tested. It is proposed that pathology in RCPm muscles has been undervalued, primarily because of their small size and a misunderstanding of their functional significance. By actively restricting the study cohort to a specific headache population, the power of the statistical analysis will be increased. It is hypothesized that the combined use of OMT and THE will decrease headache measures of frequency, intensity and duration, will increase the CSA and reduce the percentage of fatty infiltration (FI) of RCPm muscles on MRI, and will reduce forward head posture (FHP) in female patients diagnosed with CeH.

ELIGIBILITY:
Inclusion Criteria: Females diagnosed with chronic cervicogenic headache.

Exclusion Criteria:

* Have you been involved in a rear-end motor vehicle accident within the past 3 years?
* Have you had spinal surgery performed on your neck?
* Do you have a pinched nerve in the neck that produces pain radiating down your arm.
* Have you been diagnosed with diseases such as rheumatoid arthritis, lupus, or ankylosing spondylitis.
* Do you have ongoing central nervous system pathology such as hemiparesis, cervical radiculopathy, spondylolisthesis grade III or IV, central nervous system causes of balance & coordination deficits, orthostatic hypotension, vestibular disorders, pregnancy, recent spinal fractures, moderate to severe traumatic brain injury.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Cervicogenic Headache | 18 months
  Reduction of headache frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States